CLINICAL TRIAL: NCT04200378
Title: Invasive Hemodynamic Response to Transcatheter Edge-to-Edge Mitral Valve Repair
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mackram F. Eleid, Principal Investigator, Mayo Clinic
Other Study IDs: 19-004449
Record Dates: First submitted 2019-12-13; First posted 2019-12-16 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Draw
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects undergoing TMVr: Subjects with severe, symptomatic primary mitral regurgitation (MR) scheduled to undergo a transcatheter mitral valve repair (TMVr) as standard of care will have intra-op baseline and post repair blood draws. Pre-procedure and post-procedure transthoracic echocardiograms (TTE) will assess the hemodynamic implications of the repair.

SUMMARY:
Studying the effects of Trans-catheter Mitral Valve Repair (TMVr) on the hemodynamics and biomarkers in patients with severe mitral valve regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years) with severe, symptomatic primary mitral regurgitation identified by Doppler transthoracic echocardiogram
* Heart team (cardiologist and cardiac surgeon) agree that patient would be eligible for TMVR with Transcatheter edge to edge repair device.
* TMVR procedure will be performed in the cardiac catheterization laboratory for hemodynamic data recording

Exclusion Criteria:

* Women who are pregnant or believe they could be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving a standard of care TMVR with Transcatheter edge to edge repair device for mitral regurgitation symptom alleviation.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Change in stroke volume index | Baseline, approximately 10 mins after valve repair
  Change in stroke volume index 10 minutes post repair to baseline stroke volume index measurement (L/m^2)
Change in cardiac index | Baseline, approximately 10 mins after valve repair
  Change in cardiac index 10 minutes post repair to baseline cardiac index measurement (L/min/m^2)

CONTACTS AND LOCATIONS:
Overall Officials: Mackram Eleid, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials